CLINICAL TRIAL: NCT00429637
Title: Phase 2 Continuous Exhaled Breath Condensate pH in Mechanically Ventilated Patients
Brief Title: Continuous Exhaled Breath Condensate pH in Mechanically Ventilated Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Other Study IDs: 11618
Record Dates: First submitted 2007-01-30; First posted 2007-02-01 (Estimated); Last update posted 2008-08-07 (Estimated); Status verified 2008-08

CONDITIONS: Respiratory Distress Syndrome, Adult; Respiratory Syncytial Virus Infections; Pneumonia; Acute Lung Injury
Keywords: EBC pH; Airway acidification; Condensimetry; ARDS; RSV; ALI; Airway reconstruction
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Syncytial Virus Infections; Pneumonia; Acute Lung Injury

SUMMARY:
Given the possible prognostic relationship between exhaled breath condensate pH and clinical symptoms, it is quite plausible that exhaled breath condensate pH can prove useful in the intensive care unit. For example, if exhaled breath condensate pH falls prior to the onset of clinical symptoms, it is likely that it can be useful as an early marker, heralding the onset of various inflammatory lung diseases. Specifically, exhaled breath condensate pH could be used as a safe, non-invasive screening tool for Ventilator Associated Pneumonia. Similarly, just as changes in exhaled breath condensate pH might predict the onset of disease, exhaled breath condensate pH changes might also mark the progression or resolution of disease (e.g. alerting clinicians to possible readiness for extubation). Although such notions are hypothetical, they are beginning to be supported by anecdotal evidence.

DETAILED DESCRIPTION:
The investigators have developed a method of collecting exhaled breath condensate pH continually from ventilated patients, which (1) takes samples from an exhaust port on the outside of the ventilator circuit, and (2) possesses no measurable resistance to the ventilator circuit (and, therefore the sampling procedure in no way affects the patient).

Now, additionally, we have performed the continuous collection process on 10 patients in the intensive care units, none of whom have had any ill effects from the collection process.

The placement of the exhaled breath condensate collection device on the ventilator exhaust port offers a simplified, accurate, and safe method of investigating the relationships between airway pH and various pulmonary inflammatory disease processes in intubated patients of all ages.

In order to further extend our study of airway pH in intubated subjects, we believe it is necessary to obtain more frequent exhaled breath condensate pH measurements from intubated subjects. To that end, we have developed a collection system that will also measure the pH of the collected exhaled breath condensate in a fashion similar to the methodology used for thousands of assays in our laboratory and other laboratories globally. This involves deaeration of the sample to remove carbon dioxide. In the lab environment, this is performed with Argon. In the ICU setting, we will accomplish the same effect by using wall oxygen.

The continuous exhaled breath condensate pH collection and assay system consists of a condenser attached to the exhaust port of the ventilator. The condenser is kept chilled to slightly above freezing temperature by a refrigeration system commonly employed in ICU settings. The collection device stays attached to the exhalation port of the ventilator continuously, for hours to days.

Collected exhaled breath condensate is channeled into two deaeration chambers, through which wall oxygen is bubbled (total flow of 1 liter/min). In the second deaeration chamber, a micro pH electrode is inserted. This pH electrode is attached to a pH recorder that has internal memory that can record essentially an infinite number of measurements, allowing for any length duration of monitoring. This recorder has been evaluated by clinical engineering for radio frequency and other interference and is cleared for hospital use.

After measurement of pH, exhaled breath condensate is channeled into a waste chamber.

The breath condensate collection system is maintained chilled by a "hospital grade" Electri-Cool II model 767 refrigerated cooling system (or near-equivalent) that is clinically approved for use in the intensive care units. This device is approximately 30 cm on a side, and is kept on a wheeled cart out of the way of any clinical activity.

Hypothesis to be Tested: Clearly state the objectives and hypotheses and clearly define the primary and any secondary outcome measures.

1. Exhaled breath condensate pH will have greater within-hour variability in subjects with lung disease than in subjects intubated for non-pulmonary reasons.
2. Exhaled breath condensate pH will rise prior to readiness for extubation in infants and toddlers requiring mechanical ventilation for acute bronchiolitis.
3. A decline in exhaled breath condensate pH or an increase in exhaled breath condensate pH variability will predict the onset of pulmonary inflammatory processes (such as ventilator-associated pneumonia) in those who initially require mechanical ventilation for non-inflammatory reasons.

ELIGIBILITY:
Inclusion Criteria:

* Any intubated patients, aged birth to adulthood, who are on a ventilator in any University of Virginia (UVA) intensive care unit.

Exclusion Criteria:

* Control subjects may not be taking oral or inhaled steroids or have asthma, chronic obstructive pulmonary disease (COPD), cystic fibrosis, bacterial or viral pneumonitis, or adult respiratory distress syndrome (ARDS).

Min Age: 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2004-12; Study Completion 2009-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John F Hunt, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States